CLINICAL TRIAL: NCT06136858
Title: Cuirass Shell Fitting and Time to Visible Ventilation in Healthy Volunteers - an Observational Study.
Brief Title: Cuirass Fitting Study - Time for Mounting and Ventilation
Acronym: Cuirass
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jakob Friis Schmidt, Staff specialist anaesthesiology MD phD, Rigshospitalet, Denmark
Other Study IDs: The Cuirass Fitting Trial
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Airway Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy volunteers: participants of the Airway management Course in Copenhagen Denmark 2023
  Interventions: Device: Cuirass ventilation

INTERVENTIONS:
Device: Cuirass ventilation — We will fit the Cuirass Shell and start Biphasic Cuirass Ventilation on all participants.

SUMMARY:
Non-invasive biphasic cuirass ventilation (BCV) has recently been described for ENT surgery (ref 1-2). The clinical experience is however still sparse and further study is required.

The purpose of the study is to descibe 1) mounting time and fitting of the cuirass shell on voluntary participants and 2) time to visible ventilation

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the the fitting of the Cuirass shell on healthy volunteers. Even though there is growing knowledge of Cuirass ventilation in anaesthesia, (ref. 1-2) there is sparse experiences with the time required for fitting the Cuirass shell and the time to start of ventilation. This knowledge is paramount before even discussing the potential use of Cuirass ventilation in acute settings in the future.

In addition to the invitation to the Copenhagen Airway Management course in Copenhagen Denmark on 30th of November 2023, all participants have been invited an has accepted to participate in the study.

In total 60 to 65 participants will all have the Cuirass shell fitted and will be awake ventilated with Biphasic Cuirass Ventilation. All participants have given consent to being video filmed.

The study will register the time it takes to fit the Cuirass shell and the time before visible ventilation is obtained.

All participants will be in their habitual state i.e..no sedation is required since the product was originally designed for home use in awake patients.

ELIGIBILITY:
Inclusion Criteria:

* participants of the airway course

Exclusion Criteria:

* Recent surgery in thoracic or abdominal compartments
* participants with pace-maker

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population is healthy volunteers, mostly doctors, who participate in a large airway management course i Copenhagen.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
The primary end point of the study is to evaluate the number of participants who are fitted with the Cuirass shell and have visible ventilation in a two liters breathing bag within three minutes. | 15 minuttes
  Timing of the above

SECONDARY OUTCOMES:
Mean time for fitting of the cuirass shell and start of visible ventilation and fraction of participants who can be ventilated within one minute and within two minuttes | 15 minuttes
  timing of the above

OTHER OUTCOMES:
qualitative assessment | 15 minuttes
  During Cuirass ventilation did you experience discomfort on a scale from 1 to 10, Pain on a scale from 1 to10 And if Cuirass ventilation was the main driver of the partipants ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshopitalet, Copenhagen, Oesterbro, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kristensen MS, Hesselfeldt R, Schmidt JF. Improvements in cuirass ventilation for airway surgery: origins in Copenhagen on the 70th anniversary of the first intensive care unit. Br J Anaesth. 2023 Oct;131(4):644-648. doi: 10.1016/j.bja.2023.07.021. Epub 2023 Sep 4. PMID 37718095
- [Background] Kristensen MS, Hesselfeldt R, Schmidt JF. Modern cuirass ventilation for airway surgery: unlimited access to the larynx and trachea in anaesthetised patients. Br J Anaesth. 2023 Oct;131(4):e106-e109. doi: 10.1016/j.bja.2023.07.010. Epub 2023 Aug 14. No abstract available. PMID 37587006